CLINICAL TRIAL: NCT00002165
Title: Viracept Expanded Access Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Agouron Pharmaceuticals (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 259B; Study 515; AG1343 - 515
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1996-10

CONDITIONS: HIV Infections
Keywords: Acquired Immunodeficiency Syndrome; HIV Protease Inhibitors; CD4 Lymphocyte Count; Nelfinavir; Anti-HIV Agents
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Nelfinavir

INTERVENTIONS:
Drug: Nelfinavir mesylate

SUMMARY:
To make nelfinavir mesylate (Viracept) available for treatment of HIV positive patients who are unable to take the three commercially available protease inhibitors (because of failure, intolerance, or contraindication) and who have a CD4 cell count of <= 50. To obtain additional information on the safety profile of nelfinavir mesylate (Viracept).

(PER AMENDMENT 1/8/97: People now qualify for the Viracept Program if they are unable to take indinavir and/or ritonavir due to intolerance, contraindication or prior failure.)

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV infection.
* CD4 T cell count <= 100 cells/mm3.
* Failed, been intolerant of or had a contraindication to all three commercially available protease inhibitors (saquinavir, indinavir and ritonavir).

(PER AMENDMENT 1/8/97:

* People now qualify for the Viracept Program if they are unable to take indinavir and/or ritonavir due to intolerance, contraindication or prior failure.)

Exclusion Criteria

Prior Medication:

Excluded:

Prior therapy with Viracept.

Required:

* Indinavir.
* Saquinavir.
* Ritonavir.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Agouron Pharmaceuticals Inc, San Diego, California, United States

REFERENCES:
- [Background] New protease inhibitor available through expanded access. Posit Aware. 1996 Nov-Dec;7(6):7. PMID 11363981